CLINICAL TRIAL: NCT05435664
Title: The Effect of Progressive Relaxation Exercise on Fatigue in Intensive Care Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Selva Ezgi Askar, Lecturer, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HMKUASKAR-02
Record Dates: First submitted 2022-06-23; First posted 2022-06-28 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Intensive Care Nurse; Fatigue
Keywords: Fatigue; Intensive Care Nursing; Progressive Relaxation Exercises
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: Randomized controlled
Masking Description: There was no blinding due to the nature of the progressive relaxation exercise.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): During the first interview, the nurses in the intervention group were informed about PGE in a convenient and quiet room within the hospital, face-to-face and face-to-face. Afterwards, the researcher 15 minutes of application was made with the accompaniment. In order for the participants to practice at home, a voice recording containing the PGE steps voiced by the researcher in his own voice was sent to the nurses' phones. Nurses were asked to perform the PGE exercise by listening to the audio recording file for 15 minutes once a day for 4 weeks. In addition, daily reminders were made by creating a group over the WhatsApp application in order to prevent it from being forgotten. They were asked to provide feedback on their compliance with the program. At the beginning of the study, at the beginning of the study, at the 1st, 2nd, 3rd and 4th weeks (at the end of the application), the 'Fatigue Severity Scale' was administered again through face-to-face interviews.
  Interventions: Behavioral: Progressive relaxation exercise
- Control group (No Intervention): No intervention was made to the nurses in the control group. In the second and fourth weeks of the study, the "Fatigue Severity Scale" will be applied again through face-to-face interviews. At the end of the study, nurses will be informed about PGE and a voice recording will be sent to their phones from the WhatsApp application, containing the PGE steps, which the researcher voiced with her voice.

INTERVENTIONS:
Behavioral: Progressive relaxation exercise — It consists of sessions involving deep breathing and stretching and relaxing the body.
  Arms: Intervention Group

SUMMARY:
This study was planned as a randomized controlled experiment. It was aimed to examine the effect of progressive relaxation exercises applied to intensive care nurses on fatigue. The sociodemographic information of the participants will be collected with the 'Personal Information Form' and their fatigue levels with the 'Fatigue Severity Scale'. SPSS 22.0 package program will be used in the analysis of the data. p<0.05 will be considered significant.

DETAILED DESCRIPTION:
Intensive care nurses experience high levels of fatigue due to the physically and mentally demanding tasks they undertake. For example; Conditions such as prolonged seizures, difficulty sleeping, and heavy workload trigger this fatigue. One of the non-pharmacological interventions used in the management of fatigue experienced by intensive care nurses is progressive relaxation exercise (PGE). PGE involves voluntary, continuous and systematic stretching and subsequent relaxation of various muscle groups and was first described by Jacobson in 1938. The purpose of PGE is to focus attention on skeletal muscles and relax the whole body. While doing the exercise, the individual feels the difference between tension and relaxation in the muscles. Thus, when needed, it learns to relax in order to reduce the tension in the muscles. In the literature, it has been shown that PGE reduces the severity of fatigue caused by different chronic diseases. In this context, in this study, it is aimed to examine the effect of progressive relaxation exercise applied to intensive care nurses on fatigue and to contribute to the literature and to the fatigue management of nurses in line with the results obtained.

ELIGIBILITY:
Inclusion Criteria:

* Working for at least 6 months
* Having a Fatigue Severity Scale score of 2.8 and above
* Volunteer to participate in research

Exclusion Criteria:

* Having a problem that prevents breathing through the nose
* Having a diagnosis of Chronic Obstructive Pulmonary Disease (COPD) or Asthma
* Being pregnant
* Having physical and mental health problems that prevent communication
* Practicing any complementary method (relaxation exercise, yoga, etc.) during the study
* Informed about the research but willing to participate in the research

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Change in fatigue | At the beginning of the study, at weeks 1, 2, 3 and 4
  It was measured with the Fatigue Severity Scale. The fatigue severity scale is a short measurement tool consisting of nine questions developed by Krupp and used to measure the degree of fatigue in patients with multiple sclerosis. The validity and reliability of the scale Armutlu et al. and Cronbach's alpha coefficient was found to be 0.94. In the scale, individuals are asked to rate the fatigue they have felt during the past week from 1 to 7. Each section is scored between 1 (strongly disagree) and 7 (strongly agree). The total score is calculated by taking the average of nine items.

CONTACTS AND LOCATIONS:
Locations (1):
- Hatay Mustafa Kemal University Hospital, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alkan Y. Ş, Akansel N (2021). Yoğun Bakım Hemşirelerinde Yorgunluk ile İlgili Çalışmaların İncelenmesi. Hacettepe Üniversitesi Sağlık Bilimleri Fakültesi Dergisi, 8(2), 249 - 271. Doi: 10.21020/husbfd.804308
- [Background] Gok Metin Z, Karadas C, Izgu N, Ozdemir L, Demirci U. Effects of progressive muscle relaxation and mindfulness meditation on fatigue, coping styles, and quality of life in early breast cancer patients: An assessor blinded, three-arm, randomized controlled trial. Eur J Oncol Nurs. 2019 Oct;42:116-125. doi: 10.1016/j.ejon.2019.09.003. Epub 2019 Sep 6. PMID 31520865
- [Background] Kapucu S. Yılmaz Kütmeç C. (2018). Kronik hastalıklarda progresif gevşeme egzersizlerinin yararı. F.Ü.Sağ.Bil.Tıp.Derg. 32 (2), 111-114. http://www.fusabil.org
- [Background] Park ES, Yim HW, Lee KS. Progressive muscle relaxation therapy to relieve dental anxiety: a randomized controlled trial. Eur J Oral Sci. 2019 Feb;127(1):45-51. doi: 10.1111/eos.12585. Epub 2018 Nov 14. PMID 30430667
- [Background] Mander J, Blanck P, Neubauer AB, Kroger P, Fluckiger C, Lutz W, Barnow S, Bents H, Heidenreich T. Mindfulness and progressive muscle relaxation as standardized session-introduction in individual therapy: A randomized controlled trial. J Clin Psychol. 2019 Jan;75(1):21-45. doi: 10.1002/jclp.22695. Epub 2018 Oct 8. PMID 30295914
- [Derived] Askar Askar SE, Ovayolu OO, Ovayolu N. The effect of progressive relaxation exercise on fatigue level of intensive care nurses: A randomised controlled trial. Aust Crit Care. 2024 Sep;37(5):767-774. doi: 10.1016/j.aucc.2024.01.011. Epub 2024 Apr 15. PMID 38627114